CLINICAL TRIAL: NCT06673966
Title: Immunoinflammatory State Detection and Multimodal Brain Imaging and Electrophysiologic Changes in Schizophrenia
Acronym: SZIM
Status: Recruiting | Type: Observational
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Renrong Wu, professor, Central South University
Other Study IDs: Immune inflammation
Record Dates: First submitted 2024-10-30; First posted 2024-11-05 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders
Keywords: Schizophrenia; immunity; inflammation
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Mental Disorders; Inflammation | interventions — Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Individuals with schizophrenia: Inclusion Criteria:
  1. Clinical diagnosis that meets ICD-11 criteria for schizophrenia.
  2. Confirmation of the diagnosis of schizophrenia using the SCID-5-RV.
  Exclusion criteria:
  1. Clinical diagnosis or SCID-5-RV assessment confirming neurodevelopmental disorders, bipolar and related disorders, substance use disorders (excluding alcohol and tobacco).
  2. Presence of severe or acute physical illnesses, including traumatic brain injury, intracranial space-occupying or infectious diseases, acute cardiovascular diseases, acute respiratory system diseases, acute hematological disorders, autoimmune disease, etc.
  3. Presence of clearly defined genetic diseases, including tuberous sclerosis, multiple sclerosis, Kleefstra syndrome, 22q11.2 deletion syndrome, Prader-Willi syndrome, Klinefelter syndrome (47, XXY), etc.
  Interventions: Other: Regular follow-up assessments without intervention.
- Healthy volunteers: 1. No diagnosis of any mental disorder.
  2. First degree relatives without mental disorders.
  Exclusion criteria are the same as for the schizophrenia patient group.
  Interventions: Other: Cross-sectional assessment

INTERVENTIONS:
Other: Regular follow-up assessments without intervention. — Participants will receive a 3-month follow-up with clinical information, biological samples, and imaging data collected at baseline, 1st and 3rd months. The baseline assessment will include demographic information, medical history and previous medication use. At baseline and follow-up, patients' physical examination data (height, weight, waist and hip circumference, etc.), clinical symptom assessment scales (PANSS, SANS, SAPS, CDSS, CPSS, CGI, GAF, PSP, and SAS) and MCCB cognitive assessment data, blood and cerebrospinal fluid samples, MRI, and EEG data will be collected. Collection and store of blood and cerebrospinal fluid samples for routine laboratory tests and multi-omics including immunohistology, inflammation-related molecules, single-cell sequencing, extracellular vesicles, and other assays.
  Groups: Individuals with schizophrenia
Other: Cross-sectional assessment — Volunteers' physical examination data (height, weight, waist circumference, hip circumference, etc.), scale assessments (SCID, SCL-90, and CPSS) and MCCB cognitive assessment data, blood samples, MRI, and EEG data will be collected. Blood was collected and stored for exploring differences between patients and healthy individuals.
  Groups: Healthy volunteers

SUMMARY:
Schizophrenia is a severe mental illness that seriously affects the health and functioning of patients. Previous studies have found immunoinflammatory abnormalities in the blood, cerebrospinal fluid, central nervous system, and neuroimaging of people with schizophrenia, along with therapeutic effects of anti-inflammatory drugs on schizophrenia. These evidences suggest a close relationship between schizophrenia and immunity and inflammation. Therefore, we consider that the state of immune inflammation is a potential subtype classification basis for schizophrenia, and hypothesize that immune classification based on peripheral-central multidimensional data is related to patient's response to medication and cognition.

DETAILED DESCRIPTION:
This is a single-center prospective cohort study with longitudinal follow-up of patients with schizophrenia and cross-sectional data from healthy controls matched for sex and age. Participants who meet the inclusion and exclusion criteria will receive a 3-month follow-up with clinical information, biological samples, and imaging data collected at baseline, 1st and 3rd months. The aim of this project is to analyze peripheral-central immune-inflammatory performance and changes in patients with different clinical subtypes of schizophrenia through the use of scale assessments, biospecimen analysis, and imaging data. The Positive and Negative Symptom Scale (PANSS) is used to evaluate the patient's clinical status; MATRICS Consensus Cognitive Battery (MCCB) is used to assess cognition; biological samples such as blood and cerebrospinal fluid are used for multi-omics including immunohistology, inflammation-related molecules, single-cell sequencing, and extracellular vesicles; multi-modal imaging scans are used to react to the brain's structure, function, water molecule diffusion properties, and magnetization; EEG is used to react to the electrophysiological situation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis that meets ICD-11 criteria for schizophrenia.
2. Confirmation of the diagnosis of schizophrenia using the SCID-5-RV.

Exclusion Criteria:

1. Clinical diagnosis or SCID-5-RV assessment confirming neurodevelopmental disorders, bipolar and related disorders, substance use disorders (excluding alcohol and tobacco).
2. Presence of severe or acute physical illnesses, including traumatic brain injury, intracranial space-occupying or infectious diseases, acute cardiovascular diseases, acute respiratory system diseases, acute hematological disorders, autoimmune disease, etc.
3. Presence of clearly defined genetic diseases, including tuberous sclerosis, multiple sclerosis, Kleefstra syndrome, 22q11.2 deletion syndrome, Prader-Willi syndrome, Klinefelter syndrome (47, XXY), etc.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be recruited from outpatient or inpatient departments.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of clinical symptoms by PANSS | baseline, 1st month, 3rd month
  The change of PANSS at different follow up timepoint (lower score means a better outcome).
Change of the MCCB score | baseline, 1st month, 3rd month
  After assessment at each visit, evaluator convert raw scores to scale scores, then to normalized T scores. T scores of seven domains and composite score are further calculated. Compare the intergroup differences and longitudinal changes of the MCCB score between patients with schizophrenia and healthy volunteers, as well as patients with different clinical subtypes.(higher scores mean a better outcome.)
Changes of MRI | baseline, 1st month, 3rd month
  Compare the intergroup differences and longitudinal changes in brain structure, function, DTI, and QSM between patients with schizophrenia and healthy volunteers, as well as patients with different clinical subtypes.
Changes of peripheral and central inflammatory factors | baseline, 1st month, 3rd month
  Compare the levels and longitudinal changes of inflammatory factors in cerebrospinal fluid and blood between patients with schizophrenia and healthy volunteers, as well as patients with different clinical subtypes.
Changes of autoantibody | baseline, 1st month, 3rd month
  Compare the levels and longitudinal changes of autoantibody in cerebrospinal fluid and blood between patients with schizophrenia and healthy volunteers, as well as patients with different clinical subtypes.
Changes of peripheral immune cells | baseline, 1st month, 3rd month
  Compare the intergroup differences and longitudinal changes of immune cells in the blood between patients with schizophrenia, healthy volunteers, and patients with different clinical subtypes.
EEG physiological detection index | baseline, 1st month, 3rd month
  Detect resting state and task state EEG, analyze and calculate each bandwidth of the EEG (e.g. Alpha, Beta, Theta, etc.) and the functional E/I ratio of EEG power spectrum.

SECONDARY OUTCOMES:
Changes of other biological indicators | baseline, 1st month, 3rd month
  Compare the levels and longitudinal changes of other biological indicators between patients with schizophrenia and healthy volunteers, as well as patients with different clinical subtypes.
Change of clinical symptoms by Clinical Global Impression | baseline, 1st month, 3rd month
  The change of Clinical Global Impression at different follow up timepoint (lower score means a better outcome).
Change of social function by Personal and Social Performance Scale | baseline, 1st month, 3rd month
  Change of social function by Personal and Social Performance Scale, higher score means a better outcome.
Change of Body Mass Index | baseline, 1st month, 3rd month
  BMI = weight/height^2,To some extent, Body Mass Index(BMI) can represent the situation of peripheral metabolism.
Change of the level of blood lipids | baseline, 1st month, 3rd month
  Blood lipids include total cholesterol, low-density lipoprotein-cholesterol, triglyceride and high-density lipoprotein-cholesterol.
Change of waist-hip circumference | baseline, 1st month, 3rd month
  Change of waist-hip circumference,To some extent, waist-hip circumference can represent the situation of peripheral metabolism.
Changes of the level of fasting blood glucose | baseline, 1st month, 3rd month
  Changes of fasting blood glucose.
Changes of Scale for Assessment of Positive Symptoms | baseline, 1st month, 3rd month
  The change of Scale for Assessment of Positive Symptoms at different follow up timepoint (lower score means a better outcome).
Changes of Scale for Assessment of Negative Symptoms | baseline, 1st month, 3rd month
  The change of Scale for Assessment of Negative Symptoms at different follow up timepoint (lower score means a better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, the Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No